CLINICAL TRIAL: NCT04990206
Title: A Behavioral Intervention to Improve the Sleep Health of Adults With Obesity: A Feasibility and Acceptability Study
Brief Title: Improving Sleep Health in Adults With Overweight or Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Christopher Imes, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21050043
Record Dates: First submitted 2021-07-15; First posted 2021-08-04 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Sleep Disturbance; Sleep Wake Disorders; Sleep Disorder
MeSH Terms: conditions — Parasomnias; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): TranS-C
  Interventions: Behavioral: TranS-C

INTERVENTIONS:
Behavioral: TranS-C — TranS-C will be provided in eight weekly, one-on-one 50-minute sessions delivered remotely by two-way video conferencing. Each week will include goal setting and homework assignments which will be reviewed in the following session.
  The sessions will include information on sleep and circadian rhythms, behavioral change and motivation, and goal setting. The topics covered in the sessions include establishing regular sleep-wake times, learning a wind-down route, learning a wake-up routine, improving daytime functioning, correcting unhelpful sleep-related beliefs, and maintenance of behavior change.

SUMMARY:
This study will examine the feasibility and acceptability of the Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) in adults with poor sleep and excess weight. Additionally, the study will explore if TranS-C improves sleep health and cardiovascular outcomes.

DETAILED DESCRIPTION:
Aim 1 (Primary): Examine the feasibility and acceptability of TranS-C among adults with poor sleep health and excess weight.

Aim 2 (Exploratory): Explore the effect of TranS-C on the sleep health of adults with poor sleep and excess weight.

Aim 3 (Exploratory): Explore the effect of TranS-C on the cardiometabolic health of adults with poor sleep and excess weight.

ELIGIBILITY:
Inclusion Criteria:

* Currently own and regularly use a smart phone
* Body mass index >27 and ≤ 43
* Poor sleep health on one or more of the sleep health dimensions

Exclusion Criteria:

* Presence of an unstable condition requiring physician-supervised diet and exercise
* Physical limitations precluding ability to engage in moderate-intensity physical activity
* Pregnant or intention to become pregnant during study
* Current treatment for a serious mental illness
* Being a current shift worker
* Reported alcohol intake > 4 drinks/day for males and > 3 drinks/day for females
* Current participation in a formal weight loss program, loss of ≥ 5% weight in past 6 months, or current use of weight loss medication
* History of bariatric surgery
* Planned extended vacations, absences, or relocation during study
* Another member of household is a participant in the study
* Score > 32 on the Eating Habits Checklist, an eating disorder scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 6-months
  Percentage of potential participants screened in order to enroll 10 participants
Attrition rate | 6-months
  Percentage of enrolled participants completing the 8-week intervention
Completeness of questionnaire responses | 6-months
  Percentage of completed responses

SECONDARY OUTCOMES:
Change in composite sleep health score | 8-weeks (baseline to post-intervention)
  Change in composite measure of sleep health which is the sum of scores on 6 sleep dimensions. Each dimension will be dichotomized as either 'good (1)' or 'poor (0)' based on clinically and scientifically relevant rationales and added together. Score will range from 0-6 with higher scores representing better sleep health.
Change in sleep regularity | 8-weeks (baseline to post-intervention)
  Change in standard deviation of actigraphic wake time.
Change in sleep satisfaction | 8-weeks (baseline to post-intervention)
  Change in Pittsburgh Sleep Quality Index (PSQI) sleep quality item. Item score ranges from 'very good (0)' to 'very bad (3)'.
Change in alertness | 8-weeks (baseline to post-intervention)
  Change in Epworth Sleepiness Scale (ESS). Total score ranges from 0-24. Scores equal to or greater than 10 represent excessive daytime sleepiness.
Change in sleep timing | 8-weeks (baseline to post-intervention)
  Change in mean actigraphic sleep midpoint.
Change in sleep efficiency | 8-weeks (baseline to post-intervention)
  Change in mean actigraphic sleep efficiency.
Change in sleep duration | 8-weeks (baseline to post-intervention)
  Change in mean actigraphic sleep duration.
Change in body mass index | 8-weeks (baseline to post-intervention)
  Calculated by dividing weight in pounds by height in inches squared and multiplying by a conversion factor of 703. Weight will be measured a with Tanita Scale and Body Fat Analyzer. Height will be measured in with a stadiometer.
Change in systolic and diastolic blood pressure (BP) | 8-weeks (baseline to post-intervention)
  Average of two blood pressure readings at least two minutes apart.
Change in waist circumference | 8-weeks (baseline to post-intervention)
  Measured with a Gulick II measuring tape above the right iliac crest. Will include two measurements to the nearest 0.1 cm. If the two values are within 2 cm of each other, a mean with be calculated; if not, the measurements will be repeated until they are within 2 cm of each other.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Imes, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Nursing, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data sets from the proposed research may be shared.
Time Frame: Publications are complete.
Access Criteria: A Limited Dataset (LDS) may be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.